CLINICAL TRIAL: NCT01962857
Title: Effect of 4 Weeks of Shuttle Run Training on Insulin Sensitivity in Sedentary Men
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: No member of staff available for active recruitment at the moment
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Jason Gill, Reader in Exercise Metabolism, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FBLS1020
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Insulin Resistance; Obesity; Metabolic Syndrome
Keywords: Physical activity; Exercise; Insulin resistance; High intensity interval training; Fat oxidation; Fitness; Lipids; Blood pressure
MeSH Terms: conditions — Insulin Resistance; Obesity; Metabolic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): 4 week supervised high-intensity shuttle running intervention, with 3 sessions per week (12 sessions in total)
  Interventions: Behavioral: Exercise
- Control (No Intervention): No intervention - participants maintain usual lifestyle

INTERVENTIONS:
Behavioral: Exercise — 4-week supervised high intensity shuttle running intervention, 3 sessions per week (12 sessions in total)
  Arms: Exercise

SUMMARY:
A number of studies have shown that short duration, high intensity interval training can improve health-related outcomes, such as insulin sensitivity and cardiorespiratory fitness. However, these often use specialized equipment, such as cycle ergometers, which makes it difficult to roll these interventions out for wide-scale use in the general population. This study aims evaluate the effects of a high intensity shuttle running intervention on insulin sensitivity, fitness and related cardiometabolic risk factors in men who are currently inactive. Participants will be randomized into intervention (4 weeks of shuttle running) and control groups. We hypothesize that the shuttle running programme will result in improved insulin sensitivity, fitness and increased fat oxidation at rest compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* male
* 18-40 years
* undertaking < 1 hour per week of planned exercise

Exclusion Criteria:

* BMI > 35 kg/m2
* Blood pressure > 160/90 mm Hg (on anti-hypertensive medication)
* history of established coronary heart disease
* family history of early cardiac death (<40 years)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from baseline immediately post-intervention (4 weeks after baseline)
  Assessed from glucose and insulin concentrations in fasted state and during oral glucose tolerance test.

SECONDARY OUTCOMES:
Resting substrate utilization | Change from baseline immediately post-intervention (4 weeks after baseline)
  Metabolic rate and fat and carbohydrate oxidation estimated via indirect calorimetry
Endurance exercise performance | Change from baseline immediately post-intervention (4 weeks after baseline)
  Time taken to complete 100 x 10m shuttle runs
Sprint exercise performance | Change from baseline immediately post-intervention (4 weeks after baseline)
  Time taken to complete 10 x 10m shuttle runs
Body weight | Change from baseline immediately post-intervention (4 weeks after baseline)
Waist circumference | Change from baseline immediately post-intervention (4 weeks after baseline)
Percentage body fat | Change from baseline immediately post-intervention (4 weeks after baseline)
Clustered Cardiometabolic Risk Score | Change from baseline immediately post-intervention (4 weeks after baseline)
  Clustered Cardiometabolic Risk Score = -zHDL+zInsulin+zGlucose+zTriglycerides+( zBMI+zWC)/2+(zSBP+zDBP)/2.

OTHER OUTCOMES:
Objectively measured physical activity | Change from baseline to week 4 of intervention
  Time spent sedentary and physically active assessed by accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom